CLINICAL TRIAL: NCT06070844
Title: The Effect of Yoga Nidra on Pain, Mobility, First Walking Distance and Maternal Satisfaction After Caesarean Section
Brief Title: Yoga Nidra and Pain After Caesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aysegul Kilicli (Other)
Responsible Party: Sponsor-Investigator, Aysegul Kilicli, Gaziantep University Health Sciences Institute, Department of Nursing, Department of Obstetrics and Gynaecology Nursing, PhD., University of Gaziantep
Organization: University of Gaziantep (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: yoga nidra and caesarean
Record Dates: First submitted 2023-09-18; First posted 2023-10-06 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Caesarean Section; Yoga
Keywords: caesarean section; yoga nidra; pain; mobilization
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: randomised controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- yoga nidra (Experimental): yoga nidra
  Interventions: Behavioral: yoga nidra
- control (No Intervention): control group

INTERVENTIONS:
Behavioral: yoga nidra — Yoga Nidra is a guided meditation technique that involves listening to audio readings. Yoga nidra application will be started at the 6th postoperative hour and will be applied one time. Yoga nidra is expressed as yoga sleep or deep relaxation. In this practice, it will be ensured that the mother will mentally visualise all parts of her body with the commands to be given during controlled breathing and emotionally feel the body parts. The Yoga Nidra application will last 30 minutes.
  Arms: yoga nidra

SUMMARY:
The effect of yoga nidra on pain, mobilisation, first walking distance and maternal satisfaction after caesarean section

DETAILED DESCRIPTION:
The aim of this study is to investigate the effect of yoga nidra on pain, mobilisation, first walking distance and maternal satisfaction after caesarean section.

Sample size:

* The sample size is 128 women.
* The sample will include 64 mothers in the experimental group and 64 mothers in the control group.

Application time:

* Yoga nidra will be performed once in the sixth postoperative hour after caesarean section.
* Yoga nidra will be carried out once for each mother by the researcher Ayşegül Kılıçlı.
* The application will take 30 minutes.
* Only yoga nidra will not be applied to the control group. Other measurements and follow-ups will be carried out in parallel as in the experimental group.

Data collection tools:

* Introductory Information Form
* Visual Analogue Scale for Pain
* Patient Mobility Scale and Observer Mobility Scale
* Newcastle Satisfaction with Nursing Care Scale
* Note: Mobilisation distance will be measured with a metre.

Measurement time:

* Introductory Information Form will be filled out before application.
* Pain level will be measured immediately before the application.
* immediately after the application pain, mobilisation, first walking distance and maternal satisfaction will be measured.

ELIGIBILITY:
Inclusion Criteria:

* women who gave birth by caesarean section,
* whose birth was performed with spinal anaesthesia,
* who are 19 years of age or older and 35 years of age or younger,
* who were born at 37 or more weeks of gestation,
* who had a singleton birth,
* who do not have chronic diseases and any complications in this pregnancy and postpartum period,
* who have not performed yoga nidra practice before will be included in the study.

Exclusion Criteria:

* those who do not meet the inclusion criteria of the study,
* who do not voluntarily participate in the study,
* those who want to voluntarily leave the study at any stage after being included in the study,
* mothers who develop any health problems in the birth and postpartum period will be excluded.

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — mothers giving birth only by caesarean section in hospital
Enrollment: 128 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Cesarean Pain | immediately before yoga nidra application
  Visual Analogue Scale for Pain; It scores between 0 and 10, and the higher the score, the greater the pain.
Cesarean Pain | immediately after yoga nidra application
  Visual Analogue Scale for Pain
Patient Mobilization | immediately after yoga nidra application
  Patient Mobility Scale; The lowest and highest score that can be obtained from each item is between 0-15, and the total score is between 0-120. An increase in scale scores for the question answers in the study indicates an increase in pain and stiffness related to activity.
Observer Mobilization | immediately after yoga nidra application
  Observer Mobility Scale; The lowest and highest score that can be obtained from each item of the scale is between 1-5, and the total score is between 4-20. An increase in the score indicates insufficient mobility.
Patient Satisfaction | immediately after yoga nidra application
  Newcastle Satisfaction with Nursing Care Scale
Walking distance | immediately after yoga nidra application
  The first walking distance of the mothers will be measured with a meter.

CONTACTS AND LOCATIONS:
Locations (1):
- Şanlıurfa training and research hospital, Sanliurfa, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No